CLINICAL TRIAL: NCT00690716
Title: A Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Safety and Efficacy of Nasal Carbon Dioxide in the Treatment of Mild Headache in Migraineurs
Brief Title: The Effect of Nasal Carbon Dioxide (CO2) in the Treatment of Mild Headache in People Who Experience Migraines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Capnia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C112
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Migraine
Keywords: Nasal CO2; Phase II; Adaptive; Randomized; Double-Blind; Placebo-Controlled; Multiple-Dose; Multi-center; Safety; Efficacy; Mild Headache; Migraineur
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Nasal CO2
  Interventions: Drug: Nasal CO2
- 2 (Placebo Comparator): Inactive Placebo
  Interventions: Drug: Inactive Placebo

INTERVENTIONS:
Drug: Nasal CO2 — Adaptive Randomization to a Dosing Regimen for Treatment of a Qualifying Headache
  Arms: 1
Drug: Inactive Placebo — Adaptive Randomization to a Dosing Regimen for Treatment of a Qualifying Headache
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety and effect of nasal carbon dioxide in the treatment of mild headaches in people who have migraines.

DETAILED DESCRIPTION:
This multi-center, adaptively randomized, double-blind, placebo-controlled trial will evaluate the efficacy and safety of a nasal, non-inhaled administration of carbon dioxide (CO2) in the treatment of mild headaches. An estimated 250 patients who meet the eligibility criteria will be enrolled into this study at approximately 15 sites to ensure that about 220 patients are randomized and complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and understand informed consent form and voluntarily consent to participate in this study by signing the IRB-approved informed consent form
* Established diagnosis of migraine with or without aura per ICHD-II (patients with a diagnosis of only menstrual migraine are not eligible)
* History of 2-8 migraine attacks per month during the 3 months prior to randomization
* Have a typical migraine which progresses from a distinct mild headache to a moderate or severe migraine
* Able to recognize a mild headache that could develop into a moderate or severe migraine

Exclusion Criteria:

* Have less than 48 hours of freedom from headache between attacks of migraine
* Have 15 or more headache days per month
* Are females who are pregnant or lactating
* Use antipsychotic or antidepressant medications (unless only for migraine prophylaxis) within 12 weeks prior to randomization and for the duration of the study
* Have a concurrent diagnosis of TMD or trigeminal neuralgia requiring treatment
* Clinically significant deviated septum, nasal polyps or other nasal condition that prevents unrestricted breathing through each nostril
* Have participated in another study with nasal CO2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2008-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who are pain-free | 2 hours post study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Roger K. Cady, MD, Study Chair — Clinvest
Locations (15):
- United States (15):
  - Capnia Investigative Site, Birmingham, Alabama
  - Capnia Investigative Site, Stanford, California
  - Capnia Investigative Site, East Hartford, Connecticut
  - Capnia Investigative Site, West Palm Beach, Florida
  - Capnia Investigative Site, Chicago, Illinois
  - Capnia Investigative Site, North Dartmouth, Massachusetts
  - Capnia Investigative Site, Wellesley Hills, Massachusetts
  - Capnia Investigative Site, Ann Arbor, Michigan
  - Capnia Investigative Site, Kalamazoo, Michigan
  - Capnia Investigative Site, Springfield, Missouri
  - Capnia Investigative Site, St Louis, Missouri
  - Capnia Investigative Site, Philadelphia, Pennsylvania
  - Capnia Investigative Site, Pittsburgh, Pennsylvania
  - Capnia Investigative Site, Nashville, Tennessee
  - Capnia Investigative Site, Seattle, Washington